CLINICAL TRIAL: NCT01114971
Title: Randomized, Double-Blinded, Active-Controlled Study to Evaluate the Intraoperative Use of Labetalol vs. Esmolol for Maintaining Hemodynamic Stability During Laparoscopic Surgery: Effect on Recovery and Postoperative Pain
Brief Title: Labetalol and Esmolol: Vital Signs and Post Operative Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Ronald Wender, Chairman, Department of Anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00019328
Record Dates: First submitted 2010-04-23; First posted 2010-05-03 (Estimated); Results first posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Laparoscopic Surgery
Keywords: Labetalol; Esmolol; Fentanyl; Anesthetic adjuvant; Ambulatory surgery; Outpatient surgery; Pain management; Hemodynamic stability; Perioperative outcomes
MeSH Terms: conditions — Agnosia | interventions — Fentanyl; Labetalol; esmolol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fentanyl (Active Comparator): Fentanyl 50 micrograms/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or Heart Rate (HR) > 80 bpm)
  Interventions: Drug: Labetalol; Drug: Esmolol
- Labetalol (Experimental): Labetalol 5 mg/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
  Interventions: Drug: Fentanyl; Drug: Esmolol
- Esmolol (Experimental): Esmolol 10 mg/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
  Interventions: Drug: Fentanyl; Drug: Labetalol

INTERVENTIONS:
Drug: Fentanyl — Fentanyl 50 micrograms/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
  Arms: Esmolol; Labetalol
Drug: Labetalol — Labetalol 5 mg/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
  Arms: Esmolol; Fentanyl
Drug: Esmolol — Esmolol 10 mg/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
  Other Names: Brevibloc
  Arms: Fentanyl; Labetalol

SUMMARY:
This study proposes to investigate the effects of labetalol or esmolol on managing the vital signs (like blood pressure and heart rate) during surgery, on pain management, and on the later recovery after surgery.

It will also assess the cost-effectiveness of Labetalol and esmolol for outpatient surgery.

DETAILED DESCRIPTION:
Finding the optimal combination of anesthetic adjuvant drugs for maintaining hemodynamic stability during surgery is a challenge (1-3). Traditionally, potent opioid analgesics like fentanyl and its newer analogs have been used for this purpose. However, use of opioid compounds is associated with well-known side effects (e.g., ventilatory depression, postoperative nausea and vomiting, constipation, ileus, bladder dysfunction, urinary retention, pruritus, drowsiness and sedation). All of these common side effects interfere with the early recovery process and contribute to a delayed resumption of normal activities (4, 5). Increasingly, non-opioid analgesics (e.g. β-blockers and local anesthetics) are being utilized as adjuvant drugs during surgery for treatment of acute hyperdynamic responses (increased catecholamine release) during surgery, as well as, facilitation of the recovery process after surgery because of their anesthetic and analgesic-sparing effects. The β-blocking drugs, esmolol and labetalol have been used as an alternative to short-acting opioid analgesics for controlling the transient, acute autonomic responses during surgery (5-8), They have been shown to reduce the anesthetic requirement during intravenous (propofol) or volatile-based anesthesia (6,7,10-13) and to decrease opioid consumption intraoperatively and in the PACU (8). They may also improve hemodynamic stability during induction and emergence from anesthesia in the perioperative and early postoperative period and facilitate the resumption of normal activities after major surgical procedures. The anesthetic and analgesic-sparing effects of β -blockers also lead to a faster emergence from anesthesia and reduce postoperative opioid side effects (e.g., PONV) (14-18). Perioperative intravenous esmolol has shown improvement in perioperative outcomes, decreases acute hemodynamic responses, reduces anesthetics and opioids use during anesthesia, facilitates a faster emergence from anesthesia, reduces intraoperative and postoperative opioid requirements, reduces side effects as such as pruritus, constipation, ileus, nausea and vomiting (PONV) and thereby shortens the hospital stay. (3, 7, 13, 18)

Local anesthetics like lidocaine possess analgesic, antihyperalgesic and anti-inflammatory properties. Perioperative intravenous lidocaine has shown improvement in perioperative outcomes in patients undergoing abdominal surgery to decrease intraoperative requirement of Inhalants/Intravenous agents, opioid consumption, postoperative pain, fatigue, nausea and vomiting scores, maintain hemodynamic stability, facilitate a more rapid recovery of gastrointestinal function, improve postoperative recovery, fast resumption of normal activities of daily living and shorten length of hospital stay, when administered as an adjuvant during surgery.(19,23-29,33)

Theoretically, it would be extremely beneficial to administer an adjuvant (to patients undergoing abdominal surgery) that is capable of effectively controlling autonomic responses during surgery, while providing a faster recovery with fewer side effects. Preliminary data suggests that the perioperative effects of systemic administration of lidocaine and esmolol is most effective in facilitating bowel recovery, decreasing opioid consumption in the intra/postoperative period, and shorten length of hospital stay with early recovery. Therefore, we designed this prospective, randomized, double-blinded, active-controlled study to test the hypothesis that systemic administration of lidocaine and esmolol in combination (vs. either drug alone) for maintenance of hemodynamic stability during surgery will result in improved postoperative outcomes for patients undergoing abdominal surgery (e.g., less pain and postoperative nausea and vomiting, and faster return of bowel function and resumption of normal activities of daily living); leading to a shorten length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo outpatient surgery procedures
* Willingness and ability to sign an informed consent document
* No allergies to anesthetic or analgesic medications
* 18 - 80 years of age
* American Society of Anesthesiologists (ASA) physical status classification I - III adults of either sex
* Women of childbearing potential must be currently practicing an acceptable form of birth control, and have a negative urine pregnancy test

Exclusion Criteria:

* Patients with known allergy, hypersensitivity or contraindications to anesthetic or analgesic medications
* Patients with clinically-significant medical conditions, such as brain, heart, kidney, endocrine, or liver diseases, peptic ulcer disease or bleeding disorders
* Pregnant or lactating women
* Subjects with a history of alcohol or drug abuse within the past 3 months
* Any other conditions or use of any medication which may interfere with the conduct of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-09-03 (Actual); Primary Completion 2014-07-30 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Wender, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fentanyl: Fentanyl 50 micrograms/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or Heart Rate (HR) > 80 bpm)
  Labetalol: Labetalol 5 mg/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
  Esmolol: Esmolol 10 mg/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
- Labetalol: Labetalol 5 mg/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
  Fentanyl: Fentanyl 50 micrograms/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
  Esmolol: Esmolol 10 mg/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
- Esmolol: Esmolol 10 mg/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
  Fentanyl: Fentanyl 50 micrograms/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
  Labetalol: Labetalol 5 mg/ml boluses will be given:
  * at the induction time
  * at the time before surgical incision, and
  * as needed to maintain hemodynamic stability during the intraoperative period (MAP within 15% of the pre-induction baseline value, and/or HR > 80 bpm)
Period: Overall Study
Arm/Group | Fentanyl | Labetalol | Esmolol
Started | 25 | 25 | 25
Completed | 25 | 25 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ALL PARTICIPANTS = 75
  PARTICIPANTS PER GROUP= 25
Groups:
- Total: Total of all reporting groups
Arm/Group | Fentanyl | Labetalol | Esmolol | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (13) | 42 (14) | 49 (11) | 46 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 15 | 57
  Male | 4 | 4 | 10 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 6 | 4 | 13
  White | 19 | 19 | 19 | 57
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: Postoperative pain will be measured at PACU using a Verbal Rating Scale (VRS) from 0 to 10 VRS is a subjective measure in which individuals verbally rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain)
Time Frame: one day
Measure: Mean (Standard Deviation); unit: Score on scale 0-10
Arm/Group | Fentanyl | Labetalol | Esmolol
Number analyzed (Participants) | 25 | 25 | 25
Score on scale 0-10 | 3.2 (2) | 3 (3) | 3.9 (2.5)

2. Secondary Outcome: Number of Participant With Opioid Consumption
Description: n=Post discharge use of opioid consumption NUMBER OF PARTICIPANTS WHO TOOK PAIN KILLER PILLS
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | Fentanyl | Labetalol | Esmolol
Number analyzed (Participants) | 25 | 25 | 25
participants | 15 | 14 | 13

3. Secondary Outcome: Postoperative Nausea and Vomiting
Description: Nausea and vomiting will be measured at PACU
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Fentanyl | Labetalol | Esmolol
Number analyzed (Participants) | 25 | 25 | 25
participants | 9 | 4 | 7

4. Secondary Outcome: Return to Feeling Normal
Description: Days to report to return to feeling normal, using follow up questionnaires
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Fentanyl | Labetalol | Esmolol
Number analyzed (Participants) | 25 | 25 | 25
Days | 11 (9) | 10 (9) | 12 (10)

5. Secondary Outcome: Patient Satisfaction Using a Verbal Rating Scale From 0 to 10
Description: Patient satisfaction using a verbal rating scale from 0 to 10 Where a VRS is a subjective measure in which individuals verbally rated their level of satisfaction on an eleven-point numerical scale. The scale is composed of 0 (excellent satisfaction) to 10
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale (0-10)
Arm/Group | Fentanyl | Labetalol | Esmolol
Number analyzed (Participants) | 25 | 25 | 25
score on a scale (0-10) | 9.1 (1.6) | 9 (1.2) | 8 (2.5)

6. Secondary Outcome: Low Appetite
Description: Participant who experienced low appetite (follow up questionnaire)
Time Frame: 1 month
Measure: Number; unit: participants
Arm/Group | Fentanyl | Labetalol | Esmolol
Number analyzed (Participants) | 25 | 25 | 25
participants | 15 | 7 | 9

ADVERSE EVENTS:
Time Frame: One month
Arm/Group | Fentanyl | Labetalol | Esmolol
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No